CLINICAL TRIAL: NCT05120843
Title: Feasibility Testing of Care Coordination and Motivational Interviewing for Women With a Recent Preterm Birth
Brief Title: Testing Feasibility of Care Coordination and Motivational Interviewing for Women With a Recent Preterm Birth
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was terminated once we had collected sufficient information to proceed with the subsequent pilot trial.
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20-017871; 1K23HD102560 (NIH)
Record Dates: First submitted 2021-09-13; First posted 2021-11-15 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Preterm Birth; Health Care Utilization; Tobacco Use; Contraceptive Usage; Depression; Weight, Birth
Keywords: Preconception care; Interconception care; Postpartum care; Preventive health care; Care coordination; Motivational Interviewing
MeSH Terms: conditions — Premature Birth; Patient Acceptance of Health Care; Tobacco Use; Contraception Behavior; Depression; Birth Weight | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Other): This intervention will combine care coordination and motivational interviewing strategies.
  Interventions: Behavioral: Care coordination and motivational interviewing

INTERVENTIONS:
Behavioral: Care coordination and motivational interviewing — Interventionist will engage participants in care planning, health education, health care navigation, screening for unmet health needs or social needs, and motivational interviewing. The final intervention is expected to be six months in duration. However during this single-arm open testing phase, some participants may receive only key components of the intervention in order to assess feasibility, reach, adoption, and fidelity of those components.

SUMMARY:
This study continues an adaptation of care coordination to address the needs of women after preterm birth. This is a small single arm open trial designed to test intervention implementation and refine the intervention before ongoing feasibility testing.

DETAILED DESCRIPTION:
Interventionists will be trained in care coordination strategies and Motivational Interviewing (MI) techniques. Following training, investigators will enroll eligible women from a postpartum unit at a single hospital, or within two weeks of birth. Investigators will assess feasibility, adoption, reach, and fidelity of the intervention and of study data collections strategies. The intervention protocol will be revised to reflect these assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Less than 45 years old
3. History of preterm birth (< 34 weeks gestational age or 34 - 36 weeks with identifiable risk factors for recurrent preterm birth which may include low preventive care utilization, tobacco use, obesity, depression or anxiety, or history of unmet contraceptive needs)
4. Intention to seek pediatric care at one of two pediatric primary care sites
5. Medicaid insurance

Exclusion Criteria:

1. History of sterilization procedure.
2. Plan to move away from the area or transfer pediatric primary care within six months of enrollment.
3. Limited English proficiency

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2023-09-23 (Actual); Study Completion 2023-09-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Data will be used to refine the protocol for further testing. There are no plans to share individual participant data.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We have included a Table for the screening and enrollment phase of the study because a major goal of the study was to assess feasibility of screening and enrollment procedures, as well as reasons for non-participation. This table, and the numbers included in this table, support calculation of Outcomes 1 - 3. In addition they provide important information about feasibility that are relevant to other research in this area.
Period: Screening and Enrollment Phase
Arm/Group | Intervention Arm
Started (Screened for eligibility) | 49
Potentially Eligible on Chart Review | 28
Approached | 28
Confirmed Eligible | 22
Consented and Enrolled | 13
Completed | 13
Not Completed | 36
Not completed — Not eligible on chart review | 21
Not completed — Not eligible on in-person screening | 6
Not completed — Too much going on during hospital stay | 3
Not completed — Perceived services not needed | 2
Not completed — Recently moved to the area | 1
Not completed — No reason given | 3
Period: Intervention Phase
Arm/Group | Intervention Arm
Started | 13
Completed | 10
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Arm
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13
Gestational age at delivery [Mean (Standard Deviation); unit: weeks] — Weeks
  weeks | 33.2 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Screening Rate (Feasibility)
Description: The study team will compare the number of potentially eligible participants to those who are screened for eligibility. The number screened will be defined as the number of people whose are reviewed to approach for enrollment. The number of potentially eligible participants will be considered the number of women with preterm births with Medicaid insurance.
Time Frame: Screening phase (Up to 1 week prior to enrollment)
Population: See Participant Flow Section. The screening rate was 100% in that we were able to review all potentially eligible participants as defined here.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 49
Participants | 49

2. Primary Outcome: Enrollment Rate (Feasibility)
Description: The study team will track the proportion of eligible women approached for enrollment who enroll in the study.
Time Frame: Screening phase (Up to one week prior to enrollment)
Population: 22 patients were confirmed eligible of which 13 were consented.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 22
Participants | 13

3. Primary Outcome: Reasons for Non-participation (Acceptability)
Description: For women who decline enrollment we will ask them, if they are willing, to provide reasons for non-participation and potential study modifications that might have encouraged them to participate. Responses will be tabulated and reviewed for potential themes.
Time Frame: Screening phase (Up to 1 week prior to enrollment)
Population: See also Participant Flow Section
Measure: Number; unit: people
Groups:
- People Who Declined Participation: This outcome involves people who declined to participate in this study
Arm/Group | Intervention Arm | People Who Declined Participation
Number analyzed (Participants) | 0 | 9
people
  Too much going on during hospital stay |  | 3
  Perceived services not needed |  | 2
  Recently moved to the area |  | 1
  No reason given |  | 3

4. Primary Outcome: Retention Rate (Feasibility)
Description: The study team will track the proportion of enrolled participants who complete the intervention and the study assessments.
Time Frame: Enrollment through six months
Population: We counted the participants who completed all study data assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 13
Participants | 9

5. Primary Outcome: Number of Completed Assessments (Feasibility)
Description: The study team will track the proportion of the baseline, 3-month, and 6-month assessments that are completed.
Time Frame: Enrollment through six months
Measure: Number; unit: Completed assessments
Units Other Than Participants: Possible assessments
Arm/Group | Intervention Arm
Number analyzed (Participants) | 13
Number analyzed (Possible assessments) | 39
Completed assessments | 31

6. Primary Outcome: Care Coordination Fidelity (Feasibility)
Description: We will assess the proportion of intervention components completed, including interventionist completion of screening tools, as well as other tasks outlined in the care plan, including focused education, navigation, and addressing barriers to care, screening.
Time Frame: Enrollment through six months
Population: Though this was a pre-specified outcome, it was not properly defined prior to starting the pilot. Because this pilot approached intervention testing by delivering different components of the intervention to different individuals, we were unable to clarify the denominator for this measure. Data was not collected for this outcome measure due to a change in intervention delivery. Data for this outcome will not be collected or reported in the future.
Arm/Group | Intervention Arm
Number analyzed (Participants) | 0

7. Primary Outcome: Motivational Interviewing (MI) Fidelity (Feasibility)
Description: OnePass is a validated tool used to evaluate MI practice and assess fidelity based on review of a single session, using 23 items to assess MI components.61 This tool yields a global score while also identifying specific areas for additional practice and training. Scores range from 1 - 7 with 5 considered a minimum for competence. Interventionists will complete at least one OnePass within a month of starting MI sessions with participants.
Time Frame: Enrollment through six months
Population: Data for this outcome measure was not collected. Motivational interviewing was planned to be recorded using the OnePass validated tool. This was a feasibility outcome measure which has since been determined to be not feasible because of unanticipated difficulty identifying appropriate conversations to record for analysis. The overall study status has been updated to 'Terminated' to reflect this absence of data. Data will not be collected or reported in the future.
Arm/Group | Intervention Arm
Number analyzed (Participants) | 0

8. Secondary Outcome: Change in Autonomy Support
Description: Autonomy support will be measured with the short form of the Health Care Climate Questionnaire (6 items, range 6 - 42, Cronbach alpha 0.82). Scores on the short form 6-item version are calculated by averaging the individual item scores. Higher average scores represent a higher level of perceived autonomy support.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 10
units on a scale | -2.5 (11.1)

9. Secondary Outcome: Change in Autonomous Motivation
Description: Autonomous motivation will be measured using the Autonomous Motivation and External Regulation scales of the Treatment Self-Regulation Questionnaire (10 items, range 7 - 70, Cronbach alpha 0.90) with a higher score indicating higher emotion regulation strategy.
Time Frame: Baseline and 6 months
Population: 7 participants provided complete data on this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 7
units on a scale | -1.1 (9.9)

10. Secondary Outcome: Count of Preventive Care Visits
Description: This will include postpartum visits, visits for contraceptive management, routine preventive care visits, and visits to follow-up on complications of pregnancy (secondary prevention). Visits will be abstracted from the health record and from interventionist records.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Intervention Arm
Number analyzed (Participants) | 13
visits | 2.2 (1.3)

11. Secondary Outcome: Proportion of Recommended Care Completed
Description: This Outcome Measure reports the average percentage of the recommended care plan completed among participants. Recommended care will be abstracted from a care plan completed within the first two weeks after enrollment. Completed care will be abstracted from the health record and from interventionist records.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Intervention Arm
Number analyzed (Participants) | 13
percentage | 73 (35)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT05120843/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/43/NCT05120843/ICF_001.pdf